CLINICAL TRIAL: NCT07026786
Title: Using Mindfulness in an Enhanced Recovery After Surgery Protocol to Support Recovery After Colorectal Surgery: A Single Center RCT Feasibility Study
Brief Title: Using Mindfulness in an Enhanced Recovery After Surgery Protocol to Support Recovery After Colorectal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: UH Connor Whole Health (Unknown)
Responsible Party: Principal Investigator, Emily Steinhagen, Associate Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20250408
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pain After Surgery; Anxiety After Surgery
Keywords: Colorectal surgery patients; Mindfulness; Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Experimental): Those in the Mindfulness Intervention group will have a 30-minute Zoom session before surgery to learn simple mindfulness exercises like deep breathing, using senses, and staying focused on the present. After surgery, these participants will receive a refresher on the mindfulness curriculum and complete daily text message check-ins. Prior to surgery and after surgery, participants will also complete questionnaires.
  Interventions: Behavioral: Mindfulness Intervention
- Standard Care (No Intervention): Participants will undergo standard of care protocols prior to and after surgery, with no specific intervention related to the study protocol. After surgery, these participants will complete daily text message check-ins. Prior to surgery and after surgery, participants will also complete questionnaires.

INTERVENTIONS:
Behavioral: Mindfulness Intervention — Those in the Mindfulness Intervention group will have a 30-minute Zoom session before surgery to learn simple mindfulness exercises like deep breathing, using senses, and staying focused on the present. After surgery, these participants will receive a refresher on the mindfulness curriculum.
  Arms: Mindfulness Intervention

SUMMARY:
This study teaches participants who are having colorectal surgery how to use mindfulness to feel calmer and manage pain better. Participants will be randomized (like a flip of a coin) into one of two groups: Mindfulness Intervention or Standard Treatment. Those in the Mindfulness group will have a 30-minute Zoom session before surgery to learn simple mindfulness exercises like deep breathing, using senses, and staying focused on the present.

On the day after surgery, participants will watch a short video review of the mindfulness exercises.

Regardless of the group assigned, participants may be asked to complete questionnaires, and some participants will be asked to complete a semi-structured interview via Zoom, about 2 weeks to 1 month after surgery. Additionally, access to the mindfulness curriculum will be provided to those not randomized to that group. Investigators will collect information such as age, surgery details, pain levels, and pain medication usage. Participants will also fill out surveys before and after surgery to assess physical and mental well-being. All personal information will be kept safe, and interviews or Zoom sessions will be deleted after notes are taken without names attached.

Participants will be in this study for about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a bowel resection and enrolled in the UH Institutional ERAS pathway
* Patients will be admitted to the inpatient hospital for at least one day postoperatively
* Aged 18 or older
* Receiving surgery at designated University Hospitals locations (Cleveland Medical Center, Ahuja, St. John's Medical Center)
* English-speaking
* Access to the internet via phone, laptop, or iPad

Exclusion Criteria:

* Surgery for palliative purposes only
* Surgery for ostomy take-down only
* Discharged on day of surgery
* History of substance use disorder
* Allergy or intolerance to all opioids
* Insufficient English proficiency
* No access to the internet outside clinical settings
* Significant visual, hearing or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who completed all mindfulness interventions as measured by study logs | Up to one year

SECONDARY OUTCOMES:
Percentage of participants who complete all study questionnaires/text message reminders as measured by study logs | Up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Emily Steinhagen, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No